CLINICAL TRIAL: NCT04249869
Title: The Effect of Traditional Chinese Medicine (VGH-AD1) on Patients With Alzheimer's Disease: A Double-blinded Randomized Placebo-controlled Cross-over Study
Brief Title: The Efficacy of Traditional Chinese Herbal Medicine for Alzheimer's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: V109C-129
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Alzheimer Disease
Keywords: Chinese Herbal Medicine; Alzheimer's disease; Complementary Medicine
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: 28 participants will be recruited from the Division of Psychiatry and Neurology in a Medical Center. They will be randomized allocated into treatment and control groups, each including 14 participants. After eight weeks of taking, there is two-weeks of wash-out period. And then two groups will be switched for another eight weeks. Post-study follow up will be 4 weeks later once the intervention end. The study duration is totally 22 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo is manufactured to have the same appearance as VGH-AD1. Both VGH-AD1 and placebo will be coded as packages A and B by the manufacturer and the codes will only be revealed after the study ends. Therefore, patients and investigators will both be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive VGH-AD1 two times per day for 8 weeks, then entry 2 weeks wash-out period. Then switch to receive the placebo for another 8 weeks. Post-follow up will be 4 weeks later.
  Interventions: Drug: VGH-AD1
- Group B (Placebo Comparator): Group B will receive placebo two times per day for 8 weeks, then entry 2 weeks wash-out period. Then switch to receive the VGH-AD1 for another 8 weeks. Post-follow up will be 4 weeks later.
  Interventions: Drug: VGH-AD1

INTERVENTIONS:
Drug: VGH-AD1 — VGH-AD1 includes Yi-gan-san 3.0g, Huan-shao-dan 1.0g, Danshen(Radix et Rhizoma Salviae Miltiorrhizae) 0.75g, Tian-ma(Rhizoma Gastrodiae) 0.75g, Gou-teng(Ramulus Uncariae Cum Uneis) 0.375g, and Ba-ji-tian(Radix Morindae Officinalis) 0.375g, two times per day, each serving a small packet of 7.5 grams of concentrated granules.

SUMMARY:
This randomized, double-blinded, placebo-controlled, crossover clinical trial aims to investigate the effect of VGH-AD1, a scientific Chinese medicine powder prescription, on patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Dementia is a chronic, progressive neurodegenerative syndrome, characterized by an abroad category of non-reversible impairment in cerebral function, making a long-term and gradual decrease in the ability to mental cognitive tasks and performance of daily activities. The World Health Organization says that 47.5 million people around the world are living with dementia. Alzheimer's disease is accounting for 60-70 percent, the most common type of dementia. According to the record from the Ministry of Health and welfare in Taiwan, the population over 65-year-old is more than 3.36 million. It is estimated that there are more than 250,000 people with mental disabilities and nearly 600,000 people with mild cognitive impairment. With the aging of the population, experts predict that the number of patients suffering from Alzheimer's disease will be up to 800,000. In 2016, a study based on the health insurance database from 1997 to 2008 in Taiwan showed that 78.2 percent of patients have received Chinese medicine treatment, such as herbal medicine and acupuncture after diagnosed as Alzheimer's disease. Therefore, this clinical trial is designed as a randomized, double-blinded, placebo-controlled, crossover clinical trial that aims to investigate the effect of VGH-AD1, traditional Chinese herbal medicine powder, on Alzheimer's disease. Participants will be randomized allocated 14 participants into each group A and B. Group A will receive VGH-AD1, while group B will receive a placebo two times per day for eight weeks. Then entry two weeks wash-out period. And then two groups will be switched for another eight weeks. Post-study follow up will be 4 weeks after the intervention end. The study duration is totally 22 weeks. All participants will be assessed by the MMSE, IADL, NPI-Q, IQCODE, GDS, QOL-AD, TCM50, which will be conducted at baseline, week 8,10,18 and 22.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 65 years old regardless of gender.
2. Under the subject's and caregiver's willing and agreement.
3. According to DSM5 (American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Arlington, VA: American Psychiatric Publishing), was diagnosis of mild to moderate Alzheimer's type dementia;
4. MMSE score between 14 and 26;
5. Under standard treatment regularly over 3 months. (Includes Acetylcholinesterase inhibitor, NMDA receptor antagonist, and antipsychotics, antidepressants, mood stabilizer, and anxiolytic agents)

Exclusion Criteria:

1. Other types of dementia, such as Frontotemporal dementia, Dementia with Lewy Bodies, Vascular Dementia, and mixed type, et al;
2. Known of other neurological diseases, cranial nervous system cancer
3. Severe liver or kidney dysfunction (alanine aminotransferase>200 IU/L, aspartate transaminase>200 IU/L or serum creatinine >2.5 mg/dl);
4. Severe cardiovascular disease (heart failure, coronary heart disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Geriatric Depression Scale (GDS) | week 0, 8, 10,18,22
  The Geriatric Depression Scale (GDS) is a 30-item self-report assessment used to identify depression in the elderly, which will be conducted at baseline, week8, 10,18 and follow-up (22 weeks).
Changes of Mini-Mental State Examination (MMSE) | week 0, 8, 10,18,22
  Global cognition will be assessed by the MMSE,which will be conducted at baseline, week8, 10,18 and follow-up (22 weeks).
Changes of Neuropsychiatric Inventory(NPI-Q) | week 0, 8, 10,18,22
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) is an informant-based instrument that measures the presence and severity of 12 Neuropsychiatric Symptoms (NPS) in patients with dementia, as well as informant distress. The NPIQ will be conducted at baseline, week 8, 10,18 and follow-up (22 weeks).
Changes of Instrumental Activities of Daily Living (IADL) | week 0, 8, 10,18,22
  The instrumental activities of daily living (IADL) contains 8 items, such as shopping, cooking, doing laundry, handling finances, using telephone, mode of transportation, responsibility for own medication and housekeeping. The IADL will be conducted baseline, week 8, 10,18 and follow-up (22 weeks).
5. Changes of The Informant Questionnaire on Cognitive Decline in the Elderly (Short-IQCODE) | week 0, 8, 10,18,22
  The Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) provides ratings of an individual's changes in everyday cognitive functions during the previous 10 years. The questionnaire contains a total 26 questions with scores 0 to 5. The item includes short-term memory, living skills, writing, house chores, and financial dealing. If the performance remains the same as 10 years ago, then rate 3. If the performance is much worsened compare 10 years ago, then rate 5; oppositely rate 1.

SECONDARY OUTCOMES:
Changes of Quality of Life-Alzheimer's Disease (QOL-AD) | week 0, 8, 10,18,22
  The Quality of Life-Alzheimer's Disease (QOL-AD) has 13-items covering physical health, energy, mood, living situations, memory, family, marriage, friends, chores, fun, money, self and life as a whole. The QOL-AD uses straightforward language for simplicity, which will be conducted at baseline, 8, 10,18 and follow-up (22 weeks).
Changes of Constitution in Chinese Medicine Questionnaire (TCM50) | week 0, 8, 10,18,22
  The Constitution in Chinese Medicine Questionnaire (TCM50) consists of 60 items to classify a person into one or more of nine Body constitution(BC) types: gentleness (8 Items), Qi-deficiency (8 Items), Yang-deficiency (7 Items), Yin-deficiency (8 Items), phlegm-wetness (8 Items), wetness-heat (6 Items), blood-stasis (7 Items), Qi-depression (7 Items), and special diathesis (7 Items). Coexistence of multiple imbalanced BC types was possible which is consistent with the TCM theories. The scoring algorithm proposed in the original CCMQ was adopted in this study. A higher score in the CCMQ BC scale indicates a higher likelihood of the specific BC type, and a score of 30 is set as threshold for case definition. The CCMQ will be conducted at baseline, 8, 10,18 and follow-up (22 weeks).
Chinese medicine adverse effect assessment | week 0, 4, 8, 10, 14, 18, 22
  In order to cautiously evaluate and monitor the safety of Chinese medicine, the adverse effect assessment form should be filled each time the subject visits.

CONTACTS AND LOCATIONS:
Overall Officials: Shinn-Jang Hwang, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 2011 Taiwan Longitudinal Study on Aging Survey Report Health Promotion Administration, Ministry of Health and Welfare 2014.
- [Background] Albert MS, Blacker D. Mild cognitive impairment and dementia. Annu Rev Clin Psychol. 2006;2:379-88. doi: 10.1146/annurev.clinpsy.1.102803.144039. PMID 17716075
- [Background] Chen TB, Yiao SY, Sun Y, Lee HJ, Yang SC, Chiu MJ, Chen TF, Lin KN, Tang LY, Lin CC, Wang PN. Comorbidity and dementia: A nationwide survey in Taiwan. PLoS One. 2017 Apr 12;12(4):e0175475. doi: 10.1371/journal.pone.0175475. eCollection 2017. PMID 28403222
- [Background] Shen CY, Jiang JG, Yang L, Wang DW, Zhu W. Anti-ageing active ingredients from herbs and nutraceuticals used in traditional Chinese medicine: pharmacological mechanisms and implications for drug discovery. Br J Pharmacol. 2017 Jun;174(11):1395-1425. doi: 10.1111/bph.13631. Epub 2016 Oct 29. PMID 27659301
- [Background] Shanthi KB, Krishnan S, Rani P. A systematic review and meta-analysis of plasma amyloid 1-42 and tau as biomarkers for Alzheimer's disease. SAGE Open Med. 2015 Aug 10;3:2050312115598250. doi: 10.1177/2050312115598250. eCollection 2015. PMID 26770797
- [Background] Shekhar S, Kumar R, Rai N, Kumar V, Singh K, Upadhyay AD, Tripathi M, Dwivedi S, Dey AB, Dey S. Estimation of Tau and Phosphorylated Tau181 in Serum of Alzheimer's Disease and Mild Cognitive Impairment Patients. PLoS One. 2016 Jul 26;11(7):e0159099. doi: 10.1371/journal.pone.0159099. eCollection 2016. PMID 27459603
- [Background] Zhang A, Sun H, Wang P, Han Y, Wang X. Future perspectives of personalized medicine in traditional Chinese medicine: a systems biology approach. Complement Ther Med. 2012 Feb-Apr;20(1-2):93-9. doi: 10.1016/j.ctim.2011.10.007. Epub 2011 Nov 30. PMID 22305254
- [Background] Li L, Zhang L, Yang CC. Multi-Target Strategy and Experimental Studies of Traditional Chinese Medicine for Alzheimer's Disease Therapy. Curr Top Med Chem. 2016;16(5):537-48. doi: 10.2174/1568026615666150813144003. PMID 26268330
- [Background] Lin SK, Yan SH, Lai JN, Tsai TH. Patterns of Chinese medicine use in prescriptions for treating Alzheimer's disease in Taiwan. Chin Med. 2016 Mar 28;11:12. doi: 10.1186/s13020-016-0086-9. eCollection 2016. PMID 27028311
- [Background] Chen KH, Yeh MH, Livneh H, Chen BC, Lin IH, Lu MC, Tsai TY, Yeh CC. Association of traditional Chinese medicine therapy and the risk of dementia in patients with hypertension: a nationwide population-based cohort study. BMC Complement Altern Med. 2017 Mar 29;17(1):178. doi: 10.1186/s12906-017-1677-4. PMID 28356117
- [Background] Ho YS, So KF, Chang RC. Drug discovery from Chinese medicine against neurodegeneration in Alzheimer's and vascular dementia. Chin Med. 2011 Apr 22;6:15. doi: 10.1186/1749-8546-6-15. PMID 21513513
- [Background] Chen D, Yang X, Yang J, Lai G, Yong T, Tang X, Shuai O, Zhou G, Xie Y, Wu Q. Prebiotic Effect of Fructooligosaccharides from Morinda officinalis on Alzheimer's Disease in Rodent Models by Targeting the Microbiota-Gut-Brain Axis. Front Aging Neurosci. 2017 Dec 8;9:403. doi: 10.3389/fnagi.2017.00403. eCollection 2017. PMID 29276488
- [Background] Ma X, Tan C, Zhu D, Gang DR, Xiao P. Huperzine A from Huperzia species--an ethnopharmacolgical review. J Ethnopharmacol. 2007 Aug 15;113(1):15-34. doi: 10.1016/j.jep.2007.05.030. Epub 2007 Jun 2. PMID 17644292
- [Background] Iwasaki K, Satoh-Nakagawa T, Maruyama M, Monma Y, Nemoto M, Tomita N, Tanji H, Fujiwara H, Seki T, Fujii M, Arai H, Sasaki H. A randomized, observer-blind, controlled trial of the traditional Chinese medicine Yi-Gan San for improvement of behavioral and psychological symptoms and activities of daily living in dementia patients. J Clin Psychiatry. 2005 Feb;66(2):248-52. doi: 10.4088/jcp.v66n0214. PMID 15705012
- [Background] Mizukami K, Asada T, Kinoshita T, Tanaka K, Sonohara K, Nakai R, Yamaguchi K, Hanyu H, Kanaya K, Takao T, Okada M, Kudo S, Kotoku H, Iwakiri M, Kurita H, Miyamura T, Kawasaki Y, Omori K, Shiozaki K, Odawara T, Suzuki T, Yamada S, Nakamura Y, Toba K. A randomized cross-over study of a traditional Japanese medicine (kampo), yokukansan, in the treatment of the behavioural and psychological symptoms of dementia. Int J Neuropsychopharmacol. 2009 Mar;12(2):191-9. doi: 10.1017/S146114570800970X. Epub 2008 Dec 11. PMID 19079814
- [Background] Kawakami Z, Kanno H, Ueki T, Terawaki K, Tabuchi M, Ikarashi Y, Kase Y. Neuroprotective effects of yokukansan, a traditional Japanese medicine, on glutamate-mediated excitotoxicity in cultured cells. Neuroscience. 2009 Apr 10;159(4):1397-407. doi: 10.1016/j.neuroscience.2009.02.004. Epub 2009 Feb 7. PMID 19409210
- [Background] Egashira N, Iwasaki K, Ishibashi A, Hayakawa K, Okuno R, Abe M, Uchida N, Mishima K, Takasaki K, Nishimura R, Oishi R, Fujiwara M. Repeated administration of Yokukansan inhibits DOI-induced head-twitch response and decreases expression of 5-hydroxytryptamine (5-HT)2A receptors in the prefrontal cortex. Prog Neuropsychopharmacol Biol Psychiatry. 2008 Aug 1;32(6):1516-20. doi: 10.1016/j.pnpbp.2008.05.010. Epub 2008 May 20. PMID 18558456
- [Background] Bounda GA, Feng YU. Review of clinical studies of Polygonum multiflorum Thunb. and its isolated bioactive compounds. Pharmacognosy Res. 2015 Jul-Sep;7(3):225-36. doi: 10.4103/0974-8490.157957. PMID 26130933
- [Background] Buchter C, Zhao L, Havermann S, Honnen S, Fritz G, Proksch P, Watjen W. TSG (2,3,5,4'-Tetrahydroxystilbene-2-O- beta -D-glucoside) from the Chinese Herb Polygonum multiflorum Increases Life Span and Stress Resistance of Caenorhabditis elegans. Oxid Med Cell Longev. 2015;2015:124357. doi: 10.1155/2015/124357. Epub 2015 May 5. PMID 26075030
- [Background] Park SY, Jin ML, Chae SY, Ko MJ, Choi YH, Park G, Choi YW. Novel compound from Polygonum multiflorum inhibits inflammatory response in LPS-stimulated microglia by upregulating AMPK/Nrf2 pathways. Neurochem Int. 2016 Nov;100:21-29. doi: 10.1016/j.neuint.2016.08.006. Epub 2016 Aug 19. PMID 27545975
- [Background] Mazure CM, Swendsen J. Sex differences in Alzheimer's disease and other dementias. Lancet Neurol. 2016 Apr;15(5):451-2. doi: 10.1016/S1474-4422(16)00067-3. No abstract available. PMID 26987699
- [Background] Au B, Dale-McGrath S, Tierney MC. Sex differences in the prevalence and incidence of mild cognitive impairment: A meta-analysis. Ageing Res Rev. 2017 May;35:176-199. doi: 10.1016/j.arr.2016.09.005. Epub 2016 Oct 19. PMID 27771474